CLINICAL TRIAL: NCT07120035
Title: Examining Associations Between Fruit and Vegetable Intake, Skin Carotenoids, and Inflammation Among Racially and Ethnically Diverse Participants
Brief Title: Lycopene-rich Juice Intervention to Reduce Inflammatory Markers Among Adults With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Baylor College of Medicine (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMCIRB 23-002535
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Markers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lycopene-rich juice group (Experimental)
  Interventions: Dietary Supplement: Lycopene-rich juice

INTERVENTIONS:
Dietary Supplement: Lycopene-rich juice — We sought to deliver 8400 µg of lycopene per day, and so participants were asked to drink approximately 4 fluid ounces per day of the tomato-based, lycopene-rich juice.

SUMMARY:
The purpose of this research is to see whether a finger scanning device can accurately measure carotenoids, the colorful substances in fruits and vegetables, in people's skin. Participants are being invited to take part in this research because they are over the age of 18 years, and a healthy volunteer. To be eligible, participants must be: Non-Hispanic African American/Black, Asian, non-Hispanic White, or Hispanic/Latinx; Over 18 years of age; Able to speak, read, and understand English; Willing and able to drive to the research office, have a small amount of blood drawn by a trained phlebotomist, complete a questionnaire about health, demographics, and food consumption, have height, weight, body fat, and skin tone measured, and have skin carotenoids measured using the Veggie Meter; Willing to maintain usual levels of exercise and diet; Willing to consume juice daily for the study duration, 3 weeks. The juice will be provided to participants.

DETAILED DESCRIPTION:
Participants will be asked to drink a lycopene-rich (tomato-based) juice daily for three weeks. At each of 2 clinic visits, participants will be asked to: Fast for 10 hours before coming to the visit; BMI verification; blood draw by a trained phlebotomist to assess the carotenoids in blood and compare those with the carotenoids in skin and self-reported diet; Have weight, height, and body fat percentage measured; Have skin carotenoids measured using the Veggie Meter and skin color/melanin index measured using a skin spectrophotometer. This involves surface coloration scans of the finger and forearm; Complete demographic and diet history questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic African American/Black, Asian, non-Hispanic White, or Hispanic/Latinx
* Over 18 years of age
* Able to speak, read, and understand English
* Willing and able to drive to the research office, have a small amount of blood drawn by a trained phlebotomist, complete a questionnaire about health, demographics, and your food consumption, have height, weight, body fat, and skin tone measured, and have your skin carotenoids measured using the Veggie Meter.
* Willing to maintain your usual levels of exercise and diet.
* Willing to consume juice daily for the study duration, 3 weeks. We will provide this juice to you.

Exclusion Criteria:

* Not one of the racial/ethnic groups specified
* Under 18 years of age
* Not able to speak, read, and understand English
* Not willing to drink the test juice daily
* Unable to get to the research office for the baseline and follow-up measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Plasma Carotenoids | 3 weeks
  µg/dL
Skin Carotenoid Status | 3 weeks
  Measured as skin carotenoid concentrations using the Veggie Meter which uses reflection spectroscopy.
Inflammatory Markers | 3 weeks
  Mean Fluorescence Intensity (MFI)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Pitts, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina Diabetes and Obesity Institute, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share participant data with other researchers as long as they have institutional review board approval.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD will be available to other researchers whenever they have completed ethics board (IRB) approval from their home institution.